CLINICAL TRIAL: NCT02909023
Title: Performance of the Hepatitis B Virus (HBV) ELISPOT in the Detection of the T Cellular Immune Response in Patients Infected by HBV or Cured
Brief Title: Performance of the HBV ELISPOT in the Detection of the T Cellular Immune Response in Patients Infected by HBV or Cured
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0679
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: Hepatitis B Virus; Elispot test; T cellular immune response
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis B infected patients or cured: blood samples are performed to measure active T cellular immune response during a routine visit
  Interventions: Biological: blood samples are performed to measure active T cellular immune response during a routine visit

INTERVENTIONS:
Biological: blood samples are performed to measure active T cellular immune response during a routine visit — During the visit 1 (V1), after signing the informed consent, 40 mL blood sampling are carried out and analyzed with the test ELISPOT to check if the patient shows a T immune response against HBV.
  The visit 2 will be performed 4-8 weeks (depending on the availability of the patient) following V1 visit, in case the patient shows an immune response against HBV positive T following the sample taken at V1. 150 ml blood sampling are carried out at this visit.

SUMMARY:
Activation of the immune system against a pathogen can be considered one of the most effective interventions in the field of infectious diseases.

Transgene is developing a therapeutic vaccine "TG1050" for the treatment of patients with chronic and treated Hepatitis B. This biotherapy compound is for the development of T cellular immune response in these patients in order to achieve the total elimination of infected cells.

Therefore it is necessary to have measures of ways to assess accurately and reliably the presence of such a response in the study subjects.

ELIGIBILITY:
Inclusion Criteria:

Man or woman aged ≥18 years old.

Patients with chronic hepatitis B regardless of the genotype.

* treated with nucleotide analogs approved for the treatment of hepatitis B.
* or untreated.
* with a positive or negative antigen HBe
* regardless of the level of transaminases.

Patients with a history of HBV infection (recovered) with seroconversion of antigen HBs spontaneously or under treatment.

Patient with a general state ranging 0 or 1 on the ECOG scale (Eastern Cooperative Oncology Group)

Patient who signed the informed consent

Patient with a social security affiliation

Exclusion Criteria:

patients co-infected with human immunodeficiency virus (HIV) or Hepatitis C virus (HCV).

Patients treated with interferon, immunosuppressive, or experimental treatment consisting of an unapproved molecule for the treatment of hepatitis B.

Patient unable to meet the constraints of the study

Patient transplanted

Patient with a history of cancer or autoimmune disease within 5 years

Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis B infected patients or cured
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measurement of T cell response by hepatitis B antigen detected in at least one subject. | at day 1
  The method is based on the ELISPOT test. The method measures the cytokine secretion associated with immune activation after stimulation of peripheral blood mononuclear cells

SECONDARY OUTCOMES:
The probability of detection of a positive T cell response in a single measurement | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Zoulim, PU PH, Principal Investigator — Hôpital de la Croix-Rousse
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France